CLINICAL TRIAL: NCT00078078
Title: Clinical and Basic Investigations of Methylmalonic Acidemia (MMA) and Related Disorders
Brief Title: Clinical and Laboratory Study of Methylmalonic Acidemia
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040127; 04-HG-0127
Record Dates: First submitted 2004-02-18; First posted 2004-02-19 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12-05

CONDITIONS: Organic Acidemia; Methylmalonic Acidemia; Inborn Errors of Metabolism
Keywords: Organic Acidemia; Cobalamin; Vitamin B12; Methylmalonic Acidemia; Hyperhomocysteinemia; Natural History; MMA; Metabolic Disease
MeSH Terms: conditions — Methylmalonic acidemia; Metabolism, Inborn Errors; Hyperhomocysteinemia; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Methylmalonic Acidemia: Individuals with methylmalonic acidemia

SUMMARY:
Methylmalonic acidemia (MMA), one of the most common inborn errors of organic acid metabolism, is heterogeneous in etiology and clinical manifestations. Affected patients with cblA, cblB and mut classes of MMA are medically fragile and can suffer from complications such as metabolic stroke or infarction of the basal ganglia, pancreatitis, end stage renal failure, growth impairment, osteoporosis, and developmental delay. The frequency of these complications and their precipitants remain undefined. Furthermore, current treatment protocol outcomes have continued to demonstrate substantial morbidity and mortality in the patient population. Increasingly, solid organ transplantation (liver, and/or kidney) has been used to treat patients. Disordered transport and intracellular metabolism of vitamin B12 produces a distinct group of disorders that feature methylmalonic acidemia as well as (hyper)homocysteinemia. These conditions are named after the corresponding cellular complementation class - (cblC, cblD, cblF, cblJ and cblX) - and are also heterogenous, clinically and biochemically. The genetic disorders underlying cblE and cblG feature an isolated impairment of the activity of methionine synthase, a critical enzyme involved in the conversion of homocysteine to methionine and these disorders feature (hyper)homocysteinemia. Lastly, a group of patients can have increased methylmalonic acid and/or homocysteine in the blood or urine caused by variant(s) in recently identified (ACSF3) and unknown genes.

In this protocol, we will clinically evaluate patients with methylmalonic acidemia and cobalamin metabolic defects. Routine inpatient admissions will last up to 4-5 days and involve urine collection, blood drawing, ophthalmological examination, radiological procedures, MRI/MRS, skin biopsies in some, and developmental testing. In a subset of patients who have or will receive renal, hepato- or hepato-renal transplants or have an unusual variant or clinical course and have MMA, a lumbar puncture to examine CSF metabolites will be performed. In this small group of patients, CSF metabolite monitoring may be used to adjust therapy.

The study objectives will be to further delineate the spectrum of phenotypes and characterize the natural history of these enzymopathies, query for genotype/enzymatic/phenotype correlations, search for new genetic causes of methylmalonic acidemia and/or homocysteinemia, identify new disease biomarkers and define clinical outcome parameters for future clinical trials.

The population will consist of participants previously evaluated at NIH, physician referrals, and families directed to the study from clinicaltrials.gov as well as the Organic Acidemia Association, Homocystinuria Network America and other national and international support groups. Most participants will be evaluated only at the NIH Clinical Center. However, if the NIH team decides that a patient under the age of 2 years is a candidate subject for this research protocol, that patient may enroll at the Children's National Medical Center (CNMC) site, pending approval by Dr Chapman, the Principal Investigator of the CNMC location Individuals may also enroll in the tissue collection only part of the study at the UPMC Children's Hospital of Pittsburgh or share medical history and clinical data via telemedicine visits remotely. Outcome measures will largely be descriptive and encompass correlations between clinical, biochemical and molecular parameters.

DETAILED DESCRIPTION:
Methylmalonic acidemia (MMA), one of the most common inborn errors of organic acid metabolism, is heterogeneous in etiology and clinical manifestations. Affected patients with mut, cblA, and cblB classes of MMA are medically fragile and can suffer from complications such as metabolic stroke or infarction of the basal ganglia, pancreatitis, end stage renal failure, growth impairment, osteoporosis, and developmental delay. The frequency of these complications and their precipitants remain undefined. Furthermore, current outcomes have continued to demonstrate substantial morbidity and mortality in the patient population. Increasingly, solid organ transplantation (liver, and/or kidney) has been used to treat patients. Disordered transport and intracellular metabolism of vitamin B12 produces a distinct group of disorders that feature methylmalonic acidemia as well as (hyper)homocysteinemia. These conditions are named after the corresponding cellular complementation class - (cblC, cblD, cblF, cblJ and cblX) - and are also heterogeneous, clinically and biochemically. The genetic disorders underlying cblE and cblG feature an isolated impairment of the activity of methionine synthase, a critical enzyme involved in the conversion of homocysteine to methionine and these disorders feature (hyper)homocysteinemia. Lastly, a group of patients can have increased methylmalonic acid and/or homocysteine and/or malonic acid in the blood or urine caused by variant(s) in recently identified (ACSF3) and unknown genes.

In this protocol, we will clinically evaluate patients with methylmalonic acidemia and cobalamin metabolic defects. Routine inpatient admissions and outpatient evaluations will last up to 4-5 days and involve urine collection, blood drawing, ophthalmological examination, radiological procedures, MRI/MRS, skin biopsies in some, and developmental testing.

The study objectives will be to further delineate the spectrum of phenotypes and characterize the natural history of these enzymopathies, query for genotype/enzymatic/phenotype correlations, search for new genetic causes of methylmalonic acidemia and/or homocysteinemia, identify new disease biomarkers and define clinical outcome parameters for future clinical trials. The population will consist of participants previously evaluated at NIH, physician referrals, and families directed to the study from clinicaltrials.gov as well as the Organic Acidemia Association, Homocystinuria Network America and other national and international support groups. Most participants will be evaluated only at the NIH Clinical Center. However, if the NIH team decides that a patient under the age of 2 years is a candidate subject for this research protocol, that patient may enroll at the Children s National Medical Center (CNMC) site, pending approval by Dr. Chapman, the Principal Investigator of the CNMC location. Individuals may also enroll in the tissue collection only part of the study at the UPMC Children s Hospital of Pittsburgh or share medical history and clinical data via telemedicine visits remotely. Outcome measures will largely be descriptive and encompass correlations between clinical, biochemical and molecular parameters.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients of any sex, ethnicity, and over 1 month of age with biochemical or genetic diagnosis of methylmalonic acidemia or cobalamin disorders are eligible to enroll in this protocol. The primary reason for expanding enrollment to young children is because individuals with cobalamin C deficiency (cblC) develop a maculopathy often in utero or early infancy yet the natural history of the disease progression in these early years has not been well defined. Our colleagues at the National Eye Institute have documented the retinal findings in the largest cohort of individuals with cblC and have developed an expertise in this disorder. A recent report suggests that early treatment may significantly improve the retinal disease and will be the focus of a future clinical trial at the NIH Clinical Center requiring a need for more natural history data from birth to early childhood. Children ages 1 month to 2 years or under 12 kg will be reviewed by the Pediatric Consult Service prior to scheduling and if approved will be evaluated in the outpatient clinic for limited evaluations blood draw, eye exam, consults. Affected infants that are not approved by the Pediatric Consult Service or are not stable enough to travel may enroll remotely by telemedicine to include in natural history data collection, such as medical history and laboratory result sharing and interpretation, molecular genetic testing, genetic counseling, nutrition consult with dietary food log analysis, neurocognitive assessments. Affected individuals of any of the other disorders under study, younger than 2 years may be evaluated at Children s National Medical Center (CNMC) as part of an evolving agreement in the Translational Program in Pediatrics, if they are deemed eligible for participation by the NIH team and the CNMC team. Patients will be diagnosed based on a determination of MMA and homocysteine levels in plasma and urine. Most will have their complementation class known or pending. Molecular genetic analyses to determine mutations will be expected to have been performed prior to acceptance into the study. Some patients who have not yet had these laboratory tests will be admitted to the protocol based upon metabolic parameters and clinical history. This latter category of patients might include individuals with a suspected genetic but unknown type of MMA.

EXCLUSION CRITERIA:

The PI/AI may decline to enroll a patient for reasons such as being medically unstable, residing in a hospital, sub-optimal metabolic control or for any concerns arising after review of the laboratory and clinical data; any patient who requires dialysis once or more/week and weighs <40 kg; any patient who is being treated for an intercurrent infection with antibiotics or has evidence of an acute infection and has metabolic symptoms; any patient who does not have a regular/local metabolic, genetic or endocrine physician and/or a family physician, pediatrician, or internist; any patient who may be metabolically unstable but not acutely ill; and any patient or family who may not be able to institute recommendations for appropriate testing and care before visiting the NIH. Each family may be contacted by the NIH team prior to a pending admission to confirm that the patient is metabolically stable and ready to visit the NIH in a state of relative health, with an adequate supply of special formulas, medications, supplements, and if needed, medical equipment such as feeding pumps and replacement parts for feeding tubes. A subset of participants will be enrolled in the tissue collection part of the study only (i.e. if they are too sick to travel).

Pregnant women may be eligible to enroll in the study if they are affected with methylmalonic acidemia or a cobalamin disorder or are family members of an affected subject. Pregnant women are not excluded because it is important to learn more about the effects of these disorders in pregnant participants and the fetus. This research involves no more than minimal risk to the fetus. Affected subjects who are pregnant or become pregnant during their participation on the study will not be withdrawn, but will be excluded from some procedures until the pregnancy is concluded. Affected subjects who are pregnant may undergo procedures as part of their clinical care, including blood draws, genetic studies, and consultations, according to the clinical judgement of the clinical team. Pregnant participants will be excluded from some procedures such as stable isotope, GFR testing, and MRI until the pregnancy is concluded.

Patients with methylmalonic acidemia or cobalamin disorders of any age, sex and ethnicity, undergoing a transplantation surgery at UPMC Children s Hospital of Pittsburgh, are eligible to participate in the tissue collection arm of the study. Pregnant women will be excluded from tissue collection at the UPMC Children s Hospital of Pittsburgh.

For the healthy volunteers, eligibility criteria include individuals that are age 18 and over.

Exclusion criteria include: women who are pregnant, individuals being treated with antibiotics, individuals with kidney or liver disease, individuals on a special diet such as a high protein diet or taking protein supplements and individuals with severe claustrophobia or other anxiety disorders.

Ages: 1 Month to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with methylmalonic acidemia
Sampling Method: Non-Probability Sample
Enrollment: 2275 (Estimated)
Dates: Start 2004-06-07 (Actual)

PRIMARY OUTCOMES:
Natural history to assess long term complications of disease | ongoing
  assessing the complications of MMA during a week long evaluation with imaging, labs and consultations

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Venditti, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Study is observational natural history study that is ongoing with no defined endpoints.

REFERENCES:
- [Background] Manoli I, Sysol JR, Epping MW, Li L, Wang C, Sloan JL, Pass A, Gagne J, Ktena YP, Li L, Trivedi NS, Ouattara B, Zerfas PM, Hoffmann V, Abu-Asab M, Tsokos MG, Kleiner DE, Garone C, Cusmano-Ozog K, Enns GM, Vernon HJ, Andersson HC, Grunewald S, Elkahloun AG, Girard CL, Schnermann J, DiMauro S, Andres-Mateos E, Vandenberghe LH, Chandler RJ, Venditti CP. FGF21 underlies a hormetic response to metabolic stress in methylmalonic acidemia. JCI Insight. 2018 Dec 6;3(23):e124351. doi: 10.1172/jci.insight.124351. PMID 30518688
- [Background] Manoli I, Myles JG, Sloan JL, Shchelochkov OA, Venditti CP. A critical reappraisal of dietary practices in methylmalonic acidemia raises concerns about the safety of medical foods. Part 1: isolated methylmalonic acidemias. Genet Med. 2016 Apr;18(4):386-95. doi: 10.1038/gim.2015.102. Epub 2015 Aug 13. PMID 26270765
- [Background] Manoli I, Sloan JL, Venditti CP. Isolated Methylmalonic Acidemia. 2005 Aug 16 [updated 2022 Sep 8]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1231/ PMID 20301409
- [Background] Manoli I, Sysol JR, Head PE, Epping MW, Gavrilova O, Crocker MK, Sloan JL, Koutsoukos SA, Wang C, Ktena YP, Mendelson S, Pass AR, Zerfas PM, Hoffmann V, Vernon HJ, Fletcher LA, Reynolds JC, Tsokos MG, Stratakis CA, Voss SD, Chen KY, Brown RJ, Hamosh A, Berry GT, Chen XS, Yanovski JA, Venditti CP. Lipodystrophy in methylmalonic acidemia associated with elevated FGF21 and abnormal methylmalonylation. JCI Insight. 2024 Feb 22;9(4):e174097. doi: 10.1172/jci.insight.174097. PMID 38271099
- [Background] Manoli I, Pass AR, Harrington EA, Sloan JL, Gagne J, McCoy S, Bell SL, Hattenbach JD, Leitner BP, Duckworth CJ, Fletcher LA, Cassimatis TM, Galarreta CI, Thurm A, Snow J, Van Ryzin C, Ferry S, Mew NA, Shchelochkov OA, Chen KY, Venditti CP. 1-13C-propionate breath testing as a surrogate endpoint to assess efficacy of liver-directed therapies in methylmalonic acidemia (MMA). Genet Med. 2021 Aug;23(8):1522-1533. doi: 10.1038/s41436-021-01143-8. Epub 2021 Apr 5. PMID 33820958
- [Background] Sloan JL, Carrillo N, Adams D, Venditti CP. Disorders of Intracellular Cobalamin Metabolism. 2008 Feb 25 [updated 2021 Dec 16]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1328/ PMID 20301503
- [Derived] Manoli I, Gebremariam A, McCoy S, Pass AR, Gagne J, Hall C, Ferry S, Van Ryzin C, Sloan JL, Sacchetti E, Catesini G, Rizzo C, Martinelli D, Spada M, Dionisi-Vici C, Venditti CP. Biomarkers to predict disease progression and therapeutic response in isolated methylmalonic acidemia. J Inherit Metab Dis. 2023 Jul;46(4):554-572. doi: 10.1002/jimd.12636. Epub 2023 Jun 6. PMID 37243446
- [Derived] Harrington EA, Sloan JL, Manoli I, Chandler RJ, Schneider M, McGuire PJ, Calcedo R, Wilson JM, Venditti CP. Neutralizing Antibodies Against Adeno-Associated Viral Capsids in Patients with mut Methylmalonic Acidemia. Hum Gene Ther. 2016 May;27(5):345-53. doi: 10.1089/hum.2015.092. Epub 2016 Mar 22. PMID 26790480
- [Derived] Caterino M, Chandler RJ, Sloan JL, Dorko K, Cusmano-Ozog K, Ingenito L, Strom SC, Imperlini E, Scolamiero E, Venditti CP, Ruoppolo M. The proteome of methylmalonic acidemia (MMA): the elucidation of altered pathways in patient livers. Mol Biosyst. 2016 Feb;12(2):566-74. doi: 10.1039/c5mb00736d. PMID 26672496
- [Derived] Ktena YP, Ramstad T, Baker EH, Sloan JL, Mannes AJ, Manoli I, Venditti CP. Propofol administration in patients with methylmalonic acidemia and intracellular cobalamin metabolism disorders: a review of theoretical concerns and clinical experiences in 28 patients. J Inherit Metab Dis. 2015 Sep;38(5):847-53. doi: 10.1007/s10545-015-9816-x. Epub 2015 May 19. PMID 25985870
- [Derived] Raval DB, Merideth M, Sloan JL, Braverman NE, Conway RL, Manoli I, Venditti CP. Methylmalonic acidemia (MMA) in pregnancy: a case series and literature review. J Inherit Metab Dis. 2015 Sep;38(5):839-46. doi: 10.1007/s10545-014-9802-8. Epub 2015 Jan 8. PMID 25567501
- [Derived] Baker EH, Sloan JL, Hauser NS, Gropman AL, Adams DR, Toro C, Manoli I, Venditti CP. MRI characteristics of globus pallidus infarcts in isolated methylmalonic acidemia. AJNR Am J Neuroradiol. 2015 Jan;36(1):194-201. doi: 10.3174/ajnr.A4087. Epub 2014 Sep 4. PMID 25190203
- [Derived] Manoli I, Sysol JR, Li L, Houillier P, Garone C, Wang C, Zerfas PM, Cusmano-Ozog K, Young S, Trivedi NS, Cheng J, Sloan JL, Chandler RJ, Abu-Asab M, Tsokos M, Elkahloun AG, Rosen S, Enns GM, Berry GT, Hoffmann V, DiMauro S, Schnermann J, Venditti CP. Targeting proximal tubule mitochondrial dysfunction attenuates the renal disease of methylmalonic acidemia. Proc Natl Acad Sci U S A. 2013 Aug 13;110(33):13552-7. doi: 10.1073/pnas.1302764110. Epub 2013 Jul 29. PMID 23898205
- [Derived] O'Shea CJ, Sloan JL, Wiggs EA, Pao M, Gropman A, Baker EH, Manoli I, Venditti CP, Snow J. Neurocognitive phenotype of isolated methylmalonic acidemia. Pediatrics. 2012 Jun;129(6):e1541-51. doi: 10.1542/peds.2011-1715. Epub 2012 May 21. PMID 22614770
- [Derived] Hauser NS, Manoli I, Graf JC, Sloan J, Venditti CP. Variable dietary management of methylmalonic acidemia: metabolic and energetic correlations. Am J Clin Nutr. 2011 Jan;93(1):47-56. doi: 10.3945/ajcn.110.004341. Epub 2010 Nov 3. PMID 21048060
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-HG-0127.html